CLINICAL TRIAL: NCT02137629
Title: VIDAZA® Drug Use Examination
Brief Title: Post Marketing Surveillance to Collect and Evaluate the Safety and Efficacy Information of Korean MDS Patients Treated With VIDAZA®, After Approval of Marketing Authorization for New Drug in Korea
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPMS-Celgene-KOR-001
Record Dates: First submitted 2014-02-07; First posted 2014-05-14 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic syndromes; Vidaza; Observational study; Korea
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Korean patients: All Korean patients intended to be treated with Vidaza® according to the approved package insert
  Interventions: Drug: Vidaza®

INTERVENTIONS:
Drug: Vidaza® — The recommended starting dose for the first treatment for all patients regardless of baseline hematology values is Vidaza® 75mg/m2 subcutaneous(SC) injection or intravenous (IV) infusion, daily for 7 days.

SUMMARY:
The main purpose of VIDAZA® DUE (Drug Use Examination) is to collect and evaluate the safety information of Korean MDS patients treated with VIDAZA®(SC or IV) according to the approved package insert, after approval of marketing authorization for new drug in Korea. In addition, the efficacy information of VIDAZA® in clinical practice is collected and evaluated. This DUE is a prospective, multi-centre, observational, non-interventional, post-marketing surveillance. At least 600 patients' data that is eligible for safety assessment will be collected.

VIDAZA® DUE is to investigate frequency and change of Adverse Events(AEs)

/Adverse Drug Reactions(ADRs), Serious Adverse Events(SAEs)/Serious Adverse Drug Reactions(SADRs), unexpected AE/ADR and unexpected SAE/SADR, and to scrutinize factors influencing safety & efficacy of the drug. It is necessary to examine patients' demographics and baseline characteristics, medical history, status of VIDAZA treatment, concomitant medication and evaluation of safety and final efficacy (best response) assessment.

ELIGIBILITY:
Inclusion Criteria:

* Korean male or female Myelodysplastic Syndrome patients treated with VIDAZA®(subcutaneous or intravenous) according to the approved package insert

Exclusion Criteria:

* There's no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Korean patients who are intended to be treated with VIDAZA® according to the approved package insert
Sampling Method: Non-Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2010-12-27 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

PRIMARY OUTCOMES:
Number of patients with Adverse Events (AE) | Up to 6 years
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
  An SAE is any event that:
  * is fatal or life threatening
  * results in persistent or significant disability or or incapacity;
  * requires or prolongs existing hospitalization;
  * is a congenital anomaly/birth defect in the offspring of a patient who received medication;
  * conditions not included above that may jeopardize the patient or require intervention to prevent one of the outcomes listed above.

SECONDARY OUTCOMES:
Overall Response Rate | Up to 24 weeks
  Number of patients with response (CR, PR, mCR) based on the International Working Group (IWG 2006) response criteria for Myelodysplastic Syndrome (MDS)

CONTACTS AND LOCATIONS:
Overall Officials: Miran Moon, Study Director — Clinical Research Manager, Celgene Korea
Locations (47):
- South Korea (47):
  - Hallym University Sacred Heart Hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Kosin University Gospel Hospital, Busan
  - Dong-a University Medical Center, Busan
  - Pusan National University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Dongnam Inst. of Radiological & Medical Science, Busan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Chungbuk National University Hospital, Cheongju-si
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Daegu Fatima Hospita, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Eulji University Hospital - Daejeon, Daejeon
  - Dongguk University Ilsan Hospital, Goyang
  - Inje University Ilsan Paik Hospital, Goyang
  - National Health Insurance Service Ilsan Hospital, Goyang
  - Chosun University Hospital, Gwangju
  - Dongguk University Gyeongju Hospital, Gyeongju
  - Hwasun Chonnam National University Hospital, Hwasun-gun
  - Wonkwang University Hospital, Iksan
  - Inha University Hospital, Incheon
  - Gacheon University Gil Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Inje University Seoul Paik Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Kyunghee University Medical Center, Seoul
  - Seoul Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Boramae Medical Center, Seoul
  - Chung-ang University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - The Catholic University of Korea, St. Vicent's Hospital, Suwon
  - Ajou University Medical Center, Suwon
  - Ulsan University Hospital, Ulsan